CLINICAL TRIAL: NCT01662804
Title: Phase I Study of Humanized 3F8 Monoclonal Antibody (Hu3F8) When Combined With Interleukin-2 in Patients With High-Risk Neuroblastoma and GD2-positive Solid Tumors
Brief Title: Humanized 3F8 Monoclonal Antibody (Hu3F8) When Combined With Interleukin-2 in Patients With High-Risk Neuroblastoma and GD2-positive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-116
Record Dates: First submitted 2012-08-07; First posted 2012-08-10 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Neuroblastoma
Keywords: INTERLEUKIN 2; MAB 3F8; GD2-positive tumor; 12-116
MeSH Terms: conditions — Neuroblastoma | interventions — Interleukin-2

ARMS (1):
- hu3F8 and rIL-2 (Experimental): This phase I single arm trial assesses the toxicity of escalating doses of hu3F8 (day 1 and day 8) in the presence of 6 × 10^6 U rIL-2/m^2/d x 5 days sc (day 8 through day 12). These 2 doses of hu3F8 and 5 doses of rIL-2 constitute a treatment cycle.
  Interventions: Drug: 3F8 Monoclonal Antibody Combined with Interleukin-2

INTERVENTIONS:
Drug: 3F8 Monoclonal Antibody Combined with Interleukin-2 — One cycle has 2 days of intravenous hu3F8 treatment, given about 7 days apart. rIL-2 is administered sc daily over 5 days, beginning on the second infusion of hu3F8. To limit side-effects, patients receive analgesics and antihistamines as premedications. Cycles are 21 days. Patients can have up to 4 cycles of treatment on this study within 18 months of starting hu3F8.

SUMMARY:
The purpose of this study is to find out if "humanized 3F8" (Hu3F8) when combined with interleukin-2 (rIL2) is safe for treating neuroblastoma and other cancers. A phase 1 study means the investigators are trying to find out what side effects happen when higher and higher doses of a drug are used.

The investigators want to find out what effects, good and/or bad, Hu3F8 combined with rIL2 has on cancer. The amount of Hu3F8 that patients gets will depend on when they start treatment on this study. The amount of rIL2 will be the same for all patients. The investigators also want to find out more about how Hu3F8 works and how effective it is in attacking the disease when combined with rIL2.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have either (1) a diagnosis of NB as defined by international criteria,84 i.e., histopathology (confirmed by the MSKCC Department of Pathology) or BM metastases plus high urine catecholamine levels, or (2) a tumor that is GD2-positive.

  o A non-NB tumor is defined as GD2-positive by immunostaining with m3F8. If fresh or frozen tumor is not available for immunostaining, patients will be considered eligible if published reports show that >50% of that tumor type is GD2-positive by immunohistochemistry. (Note: Tissues must be fresh/frozen as fixed, paraffin-embedded specimens are unsuitable for anti-GD2 immunostaining). Tumors known to be GD2- positive by this criteria do not need immunostaining. These include: Melanoma (>50%), Desmoplastic small round cell tumors (70%), Osteosarcoma (88%) and Soft tissue sarcomas including liposarcoma, fibrosarcoma, malignant fibrous histiocytoma, leiomyosarcoma, and spindle cell sarcoma (93%).
* Patients must have either (1) refractory or relapsed high-risk NB (including MYCN-amplified stage 2/3/4/4S of any age and MYCN-nonamplified stage 4 in patients greater than 18 months of age)resistant to standard therapy*, or (2) refractory or relapsed GD2-positive tumor after receiving available life-prolonging therapies.

  *For NB, standard therapy generally includes 5-8 cycles of high dose induction chemotherapy followed by resection of gross residual tumor, with or without myeloablative chemotherapy with peripheral blood stem cell rescue and radiation therapy to the primary site. There are also salvage chemotherapy regimens for residual disease after standard induction therapy or for relapsed NB. Some examples of these chemotherapy combinations are: high-dose cyclophosphamide, topotecan and vincristine; high-dose cyclophosphamide, irinotecan and vincristine; irinotecan and temozolomide; or ifosfamide, carboplatin and etoposide.
* Patients must be older than 1 year of age.
* Prior treatment with murine 3F8 is allowed. Patients with prior m3F8, hu3F8, ch14.18 or hu14.18 treatment must have HAHA antibody titer less than or = to 1300 Elisa units/ml
* White blood cell count ≥1000/ul
* Absolute neutrophil count ≥500/ul
* Absolute lymphocyte count ≥500/ul
* Platelet count ≥25,000/ul
* No chemotherapy or immunotherapy for a minimum of three weeks prior to study enrollment
* Women of child-bearing potential must be willing to practice an effective method of birth control while on treatment
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Existing major organ dysfunction > grade 2, with the exception of hearing loss and hematologic toxicity (defined as suppression of all subtypes of WBCs, RBCs, and platelets).
* Hematologic and primary CNS malignancies
* Active life-threatening infection.
* Pregnant women or women who are breast-feeding.
* Inability to comply with protocol requirements.

Min Age: 13 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-08-06 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dosage | 1 year
  of hu3F8 when combined with rIL-2. six dosage levels of hu3F8 will be tested with three to six patients at each dosage level.

SECONDARY OUTCOMES:
pharmacokinetics | 1 year
  of iv hu3F8 in the presence of rIL-2. Pharmacokinetics will be measured by serial blood sampling following the first two iv doses of hu3F8. Serum hu3F8 will be measured at time 0, 5 min, 3h, 6-8h, 24h, 48h, 72h, 96, 120h and 168h after infusion for each of the two hu3F8 injections during the first cycle. Peak hu3F8 level at 5 min after infusion will also be measured for all hu3F8 infusions during all other cycles. PK analysis will be carried out by noncompartmental analysis of the serum concentration-time data using the WinNonlin software program (Pharsight Corp., Mountain View, CA).
anti-tumor activity | 1 year
  of hu3F8 plus rIL-2 against NB and other GD2-positive tumors. For neuroblastoma, anti-tumor activity will be measured by international neuroblastoma response criteria (INRC).90 For other solid tumors, the response and progression will be evaluated in this study using the Response Evaluation Criteria in Solid Tumors (RECIST) Committee, version 1.1.
biologic correlates with hu3F8 dose | 1 year
  Biologic correlate studies include (1) host immunity and (2) host WBC cytolytic capacity. The parameters measured for each patient under "host immunity" include: the induction of HAMA or HAHA, the induction of Ab3, the induction of Ab3', the induction of antibody response to tumor antigen and secondary cytokine profile.
quantification of pain | 1 year
  As patient's pain will be assessed with a numerical score of 1 to 10 over the course of the treatment, a curve of pain intensity over time can be generated for each patient. We have been collecting similar pain data for patients being treated with murine 3F8 (control group) and Hu3F8 alone and may be able use this to compare to pain data of patients receiving hu3F8 and rIL2. Because the first dose of hu3F8 will be given without rIL2 and the second dose with rIL2, we will also be able to directly compare the pain associated with hu3F8 with and without rIL2 in the same patient. This pain level will be compared to the pain scores in patients receiving m3F8 on concurrent protocols at 80 mg/m2/day or 20 mg/m2/day. Differences will be tested for significance using both Mann-Whitney and repeated measures ANOVA tests as described previously.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Roberts, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/